CLINICAL TRIAL: NCT03689647
Title: Reducing Metabolic Cost of Walking by Exploiting Arm Swing to Drive Leg Swing
Brief Title: Using the Arms to Drive the Legs During Walking
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: University of Houston (Other)
Responsible Party: Principal Investigator, Christopher Arellano, Assistant Professor, University of Houston
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: STUDY00001219
Record Dates: First submitted 2018-09-27; First posted 2018-09-28 (Actual); Last update posted 2018-10-02 (Actual); Status verified 2018-09

CONDITIONS: Metabolic Cost of Walking With Arm Swing Assistive Device

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Single Group Experimental (Experimental): Each participant will act as their own control with variables of interest measured while walking without the assistive device and while walking with the assistive device.
  Interventions: Device: Arm Swing Driven Assistive Apparatus

INTERVENTIONS:
Device: Arm Swing Driven Assistive Apparatus — The investigators are testing a simple, custom built apparatus to determine if it can facilitate the use of the arms to swing the legs during walking. More specifically, the investigators will measure how this assistive apparatus affects the metabolic cost and biomechanics of walking.

SUMMARY:
This study aims to understand and compare the metabolic and mechanical demands placed on the body while walking normally and walking with the use of an apparatus that drives leg swing through the use of the arms. This information will help the investigators identify how arm swing mechanics helps minimize energy demands and to use this knowledge to design walking rehabilitation interventions in the future.

ELIGIBILITY:
Inclusion Criteria:

* Apparently healthy and free from neurological disease and/or body related injury
* Community-dwelling young men and women 18-36 yrs
* Use and be contacted by telephone
* Speak, read, understand, and complete a questionnaire in English
* Body mass index < 30 kg/m2

Exclusion Criteria:

* not of the specified age range or Body Mass Index
* inadequate aerobic fitness training
* answering "no" to question #3 on Screening Form ("Is participant in good general health?")
* answering "yes" to:
* question #4 ("any difficulty with mobility?")
* question #5 ("problems with balance/dizziness?")
* question #6 ("lingering symptoms/pain from injury?")
* question #7 ("chest pain/shortness of breath?")
* question #8 ("high blood pressure/hypertension?"), or
* questions #9, 10, 11 ("first degree family history of heart attack?")
* question #12 ("smoke cigarettes?")
* question #13 ("diabetes?")
* question #14 ("high cholesterol?")
* question #15 ("Is participant pregnant?")

Ages: 18 Years to 36 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 30 (Estimated)
Dates: Start 2018-10-01 (Estimated); Primary Completion 2018-12-31 (Estimated); Study Completion 2018-12-31 (Estimated)

PRIMARY OUTCOMES:
Metabolic Cost | Change from walking without assistive apparatus to walking with assistive apparatus. Measures of metabolic cost are completed within a 3-hour time window during a single laboratory visit.
  Change in Metabolic Cost

CONTACTS AND LOCATIONS:
Overall Officials: Christopher J Arellano, PhD, Principal Investigator — University of Houston

REFERENCES:
- [Derived] Vega D, Arellano CJ. Using a simple rope-pulley system that mechanically couples the arms, legs, and treadmill reduces the metabolic cost of walking. J Neuroeng Rehabil. 2021 Jun 7;18(1):96. doi: 10.1186/s12984-021-00887-3. PMID 34098979